CLINICAL TRIAL: NCT06025110
Title: A 12-month, Randomized, Single-blind, Placebo-controlled Exposure-response Study of TCD601 (Siplizumab) in New Onset Type 1 Diabetes Patients (STRIDE)
Brief Title: A Study of TCD601 (Siplizumab) in New Onset Type 1 Diabetes Patients
Acronym: STRIDE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study has been early terminated due to business reasons. This decision is not related to any safety, efficacy, or regulatory concerns.
Sponsor: ITB-Med LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: TCD601F201
Record Dates: First submitted 2023-08-25; First posted 2023-09-06 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TCD601 (Experimental): Administered one of three doses of TCD601 over a 12 week treatment period.
  Interventions: Biological: TCD601
- Placebo (Placebo Comparator): Placebo is administered over a 12 week treatment period.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: TCD601 — Investigational Product
  Arms: TCD601
Other: Placebo — Comparator
  Arms: Placebo

SUMMARY:
The goal of this study is to determine if treatment with TCD601 improves beta-cell function in adults recently diagnosed with type 1 diabetes compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the study requirements and provide written informed consent before any study assessment is performed
* Male or female patients ≥ 18 to 45 years of age
* A diagnosis of type 1 diabetes

Exclusion Criteria:

* Women who are pregnant, lactating, or planning on pregnancy during the study
* History of cancer
* History of heart disease
* Recent infection

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Change from baseline in beta-cell function as compared to placebo at week 52. | 52 weeks
  Assess any changes in beta-cell function at the end of the study (week 52) for patients treated with TCD601 (study drug) compared to subjects treated with placebo (the comparator).

SECONDARY OUTCOMES:
Assess the incidence and severity of adverse | 52 weeks
  Number of adverse events compared to placebo at week 52.

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Juhlin, Study Director — ITB-MED
Locations (26):
- Belgium (2):
  - UZ Brussel, Brussels
  - UZ Leuven, Leuven
- Italy (4):
  - Azienda Ospedaliero-Universitaria Renato Dulbecco, Catanzaro
  - San Raffaele Hospital, Milan
  - Luigi Sacco Hospital, Milan
  - University of Siena, Siena
- Spain (6):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona
  - Hospital General de Segovia, Segovia
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clinico Universitario de Valladolid, Valladolid
- Karolinska University Hosptial, Stockholm, Sweden
- United Kingdom (13):
  - Dorset County Hospital NHS Foundation Trust, Dorchester, Dorset
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool, Merseyside
  - University of Birmingham, Birmingham
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Ninewells Hospital, Dundee
  - St George's University Hospitals NHS Foundation Trust, London
  - Guy's and St. Thomas' NHS Foundation Trust, London
  - East Kent Hospitals University NHS Foundation Trust, Margate
  - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - Oxford University Hospitals NHS Foundation Trust, Oxford
  - Northern Care Alliance NHS Foundation Trust, Salford
  - Swansea Bay University Health Board, Swansea

IPD SHARING:
Plan to Share IPD: No